CLINICAL TRIAL: NCT01353066
Title: Multicenter Randomized Prospective Trial on the Effects of Intensive Medical Treatment of Type 2 Diabetes With and Without Roux-in-Y Gastric Bypass Surgery on Carotid Intima Media Thickness in Grade I Obesity (BMI 30,0-34,9 kg/m2)
Brief Title: Gastric Bypass Versus Best Medical Treatment on Progression of Carotid-intima Media Thickness in Type 2 Diabetes Mellitus (T2DM)
Acronym: EURDSS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Antonio M Lacy, Hospital Clínic de Barcelona
Purpose: Treatment
Other Study IDs: HCB-UOM-012011
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Atherosclerotic Cardiovascular Disease; Subclinical Disease and/or Syndrome
Keywords: Type 2 Diabetes Mellitus; BMI 30.0-34.9 kg/m2
MeSH Terms: conditions — Atherosclerosis; Diabetes Mellitus, Type 2

ARMS (2):
- Intensive Medical Treatment (Active Comparator)
  Interventions: Drug: Intensive Medical Treatment
- Intensive medical treatment (IMM)+RYGBP (Experimental)
  Interventions: Other: IMM+Roux-en-Y Gastric Bypass (RYGBP)

INTERVENTIONS:
Drug: Intensive Medical Treatment
  Arms: Intensive Medical Treatment
Other: IMM+Roux-en-Y Gastric Bypass (RYGBP)
  Arms: Intensive medical treatment (IMM)+RYGBP

SUMMARY:
Background: Type 2 Diabetes Mellitus (T2DM) is associated with an increased burden for cardiovascular disease (CVD). Multifactorial interventions are necessary to reduce the CV risk in T2DM. Bariatric surgery appears to be an alternative for the multifactorial intervention in T2DM associated with obesity. Data have shown, that clinical trial aiming at the control of CVRF in T2DM may not translate in the reduction of CV events.

Hypothesis: Intensive medical treatment (IMM) including Roux-en-Y Gastric Bypass (RYGBP) could be superior in the control of the progression of subclinical atherosclerotic disease, as evaluated by carotid ultrasound, in subjects with T2DM and a BMI between 30.0 and 34.9 kg/m2.The primary aim of the study is To compare the effects of intensive medical treatment (IMM) including Roux-en-Y Gastric Bypass (RYGBP) and IMM alone on the progression of the carotid intima media thickness (CIMT) at 24 months after entry into the trial relative to baseline.Methodology: Two-year Randomized Clinical Trial, including 240 patients

ELIGIBILITY:
Inclusion Criteria:

* Age 35 to 65 years at eligibility visit.
* Diagnosed with T2DM at least 6 months prior to enrollment, under the active care of a doctor for at least he six months prior to enrollment, and HbA 1c > 7.0 %.
* Current treatment for T2DM consisting of multiple doses of insulin with/without hypoglycemic agents or hypoglycemic agents plus basal insulin.
* Optimization of diabetes medical treatment prior to inclusion in the study would have been performed based on best medical practices.
* Body Mass Index (BMI)> 30.0 kg/m2 and <34.9 kg/m2 at eligibility visit.
* Willingness to accept random assignment to either treatment group.
* Expect to live or work within approximately one hour's traveling time from the study clinic for the duration of the two-year trial.
* Willingness to comply with the follow-up protocol and successful completion of the run-in.
* Written informed consent.

Exclusion Criteria:

* Cardiovascular event (myocardial infarction, acute coronary syndrome, coronary artery angioplasty or bypass, stroke) in the past six months.
* Current evidence of congestive heart failure (grade II or IV), angina pectoris, symptomatic peripheral vascular disease or advanced cardiovascular disease.
* History of severe hypoglycemic episodes associated with medical treatment of type 2 DM
* Cardiac stress test indicating that surgery would not be safe
* Pulmonary embolus or thrombophlebitis in the past six months.
* Cancer of any kind (except basal cell skin cancer or cancer in situ) unless documented to be disease-free for five years.
* Significant anemia or history of coagulopathy.
* Serum creatinine >1.5 mg/dl.
* Serum total bilirubin or alkaline phosphatase greater than the upper limit of normal, or ALT greater than twice the upper limit of normal.
* History of previous surgery contraindicating gastric bypass at the criteria of the surgical team.
* Gastric or duodenal ulcer in the past six months.
* History of intra-abdominal sepsis (except for uncomplicated appendicitis or diverticulitis more than six months prior to enrollment).
* Previous organ transplantation.
* Self-reported HIV-positive status, active tuberculosis, active malaria, chronic hepatitis B or C, cirrhosis, or inflammatory bowel disease.
* Currently pregnant or nursing, or planning to become pregnant in the next two years.
* History of alcohol or drug dependency (excluding caffeine and nicotine) in the past five years
* Active psychosocial or psychiatric problem that is likely to interferer with adherence to the protocol.
* Score of 17 or higher on the CES-D (depression scale).
* Current participation in a conflicting research protocol.
* Presence of any chronic or debilitating disease that would make adherence to the protocol difficult.
* 12-lead EKG indicating that surgery or intensive medical treatment would not be safe.
* Diagnosed with diabetes more than 15 years ago.
* Positive GAD antibodies

Ages: 35 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)

PRIMARY OUTCOMES:
Measurement of the progression carotid intima media thickness (CIMT) at 24 months after entry into the trial relative to baseline | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Catalonia, Spain